CLINICAL TRIAL: NCT04328402
Title: Factors Correlated With Obstructive Sleep Apnea in Children and Adolescents Diagnosed by Polysomnography: Cross-sectional Study
Brief Title: Factors Correlated With Obstructive Sleep Apnea in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, PhD, Associate Professor, School of Dentistry, Federal University of Pelotas
Other Study IDs: FUPelotas6
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: diagnostic; polysomnography; sleep architecture; obstructive sleep apnea
MeSH Terms: conditions — Disease; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents submitted to PSG in sleep laboratory: Children (1 to 11 years) and adolescents (12 to 18 years), who were referred to a sleep laboratory and submitted to full-night polysomnography due to suspicious of sleep disorders.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Polysomnography, referred to as type I, allows assessing several sleep physiologic parameters (eg, EEG, electrooculogram, electromyogram, electrocardiogram, airflow, respiratory effort, oxygen saturation), whereas audio-video recording enables to document tooth-grinding sounds and distinguishing between rhythmic masticatory muscle activity (RMMA) and orofacial and other muscular activity during sleep. The apnea and hypopnea index (AHI) is defined as the number of obstructive apneas and hypopneas per hour of sleep. Obstructive Sleep Apnea is defined in PSG when AHI≥1 and is divided into the following categories, according to severity: mild OSA (AHI 1-4.9), moderate OSA (AHI 5-9.9) and severe OSA (IAH≥10). Based on the RMMA index (number of episodes per hour of sleep), sleep bruxism is diagnosed when episodes are greater than or equal to 2 (low-frequency SB, mild bruxism) or episodes are greater than or equal to 4 (high frequency SB, severe bruxism).

SUMMARY:
Obstructive Sleep Apnea (OSA) is a severe condition of sleep respiratory disorders. It is characterized by partial (hypopnea) or total (apnea) obstruction of the upper airways, negatively affecting the general and oral health of children and adolescents. The Dentistry plays a fundamental role in OSA diagnosis and early intervention, minimizing health damage and progression of the disease into adulthood. Current scientific evidence related to OSA and associated factors, as well as the prevalence and severity of the disease in children and adolescents is still scarce and presents divergences in these age groups. A retrospective cross-sectional study will be conducted to investigate the prevalence, severity and correlation between sociodemographic, behavioral, clinical and sleep quality related factors and OSA in children and adolescents diagnosed by polysomnography (PSG), using the criteria recommended by the American Academy of Sleep Medicine (AASM). The sample will consist of individuals who answered the questionnaires, performed the PSG at the Pelotas Sleep Institute and met the study inclusion criteria.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a severe condition among sleep respiratory disorders, characterized by intermittent episodes of partial (hypopnea) or total (apnea) obstruction of the upper airways during sleep. These obstructive episodes result in hypoxemia and hypercapnia, changes in intrathoracic pressure and sleep arousals, consequently leading sleep fragmentation and a non-restorative sleep pattern.

OSA affects 1 to 4% of the world's pediatric population, with a higher incidence between 2 to 8 years old, negatively affecting the general and oral health of children and adolescents. Studies show divergences regarding the prevalence among sexes, either showing similar rates for girls and boys, or a predilection of the disease for the male sex. Although scientific evidence reports known OSAs risk factors like adenotonsilar hypertrophy and obesity, there is still divergence of which associated characteristics are present in children and adolescents.

Diagnostic criteria of OSA in this population follows the recommendations of American Academy of Sleep Medicine (AASM) through the International Classification of Sleep Disorders (ICSD-3), which determines full-night PSG as the gold standard test for the diagnosis and severity of OSA, as it promotes a quantitative and objective assessment of disturbances in breathing and sleep patterns. Although parents' report of child behavior and symptoms is essential for establishing the diagnosis of OSA, the factors evaluated in the anamnesis and clinical examination, in general, do not present adequate accuracy for the diagnosis of OSA. The use of clinical history and physical examination alone is not suitable for a definite diagnose of OSA when compared to PSG. Besides, most questionnaires used as alternative diagnostic methods do not meet the necessary criteria to be considered as acceptable tools in the identification of children and adolescents with OSA.

There is evidence in the literature regarding OSA's significant morbidity in children and adolescents, leading to cardiovascular, metabolic and neurocognitive complications, resulting in reduced quality of life. Also, OSA is associated with several craniofacial and dental changes, such as retrognathia, class II malocclusion, vertical face growth and sleep bruxism. It becomes clear the importance of the dentist in identifying factors associated with OSA in children and adolescents, this being the first step towards early and definitive diagnosis, followed by adequate treatment, to minimize the health damage in this population. Therefore, this study aims to study the risk factors correlated with OSA, the prevalence and severity of illness in children and adolescents, considering that the current scientific evidence is divergent.

A retrospective cross-sectional study will be conducted to investigate the prevalence, severity and associations between diagnosis by gold-standard PSG examination and the sociodemographic, clinical conditions, sleep quality and sleep structure of children and adolescents, following the recommended criteria by the AASM. Also, this study aims to evaluate the association of sleep bruxism (SB) and OSA. The sample will consist of participants, between 1 and 18 years, who were referred to Pelotas Sleep Institute, answered the questionnaires (self-reported or parent-reported) and performed PSG for diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

* Children (1 to 11 years) and adolescents (12 to 18 years), who were referred to a sleep laboratory
* Participants who performed polysomnography and answered questionnaires (self-reported or parent-reported) at Pelotas Sleep Institute.

Exclusion Criteria:

* Participants who present a history of syndromes, neuromuscular or neurological disorders;
* Participants whose questionnaires were not completed.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants in the child and adolescent age group, referred to the Pelotas Sleep Institute for polysomnography in the period from January 2012 to December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of Obstructive Sleep Apnea (OSA) in children and adolescents evaluated by polysomnography | day 1
  Children and adolescents will be evaluated to investigate the prevalence and severity of OSA, according to the criteria of de American Association of Sleep Medicine. Participants will be diagnosed with OSA if they present: a) self-report or parent-report of snoring or difficulty breathing during sleep; and b) one or more obstructive apneas per hour of sleep in polysomnography. The apnea-hypopnea index (AHI) was calculated as the average number of apnea-hypopnea episodes per hour of sleep. Individuals with an AHI ≥ 1 were diagnosed with OSA via PSG, and its severity was classified as mild (AHI ≥ 1 and < 5 events/h), moderate (AHI ≥ 5 and < 10 events/h), and severe OSA (AHI ≥ 10 events/h).

SECONDARY OUTCOMES:
Sociodemographic and clinical condition variables | day 1
  The following sociodemographic data will be evaluated:
  1.1 Age: participants between (1 to 11 years) will be classified as children and participants between (12 to 18 years) will be classified as adolescents; 1.2 Sex: participants will be classified as (male or female); 1.3 Parental education: participants will be classified according to their parental education (< 8 years or ≥ 8 years); 1.4 Family structure: participants will be classified according to their family structure as (nuclear or non-nuclear).
  The following clinical condition data will be evaluated:
  1.5 Body mass index (BMI). Weight and height will be combined to report BMI in kg/m^2): children and adolescents will be classified as obese/ overweight/underweight/ (≥ 95th percentile/ 85th to < 95th percentile/< 5th percentile, respectively) or normal weight (5th to < 85th percentile), according to World Health Organization Child Growth Standards.
Sleep quality variables | day 1
  Sleep Quality will be evaluated with the following questions:
  1. Bedtime: how many hours does your child sleep (<8 hours or ≥8 hours); how long does it take to sleep (up to 15min, or >15 min); child resists going to bed at bedtime (no or yes); child feels anxiety or fear at bedtime (no or yes);
  2. Sleep behavior: child wakes up more than twice during the night (no or yes); child is restless and moves a lot during sleep (no or yes); child has suffocation or difficulty breathing during the night (no or yes); child sweats a lot during the night (no or yes); child grit his/her teeth while sleeping (no or yes); child has nightmares (no or yes); child snores during the night (no or yes) child has sleep enuresis (no or yes);
  3. Morning wake up: child has difficulty waking up (no or yes); child feels tired after waking up (no or yes); child is sleepy during the day (no or yes); child has headache in the morning (no or yes); child has mouth breathing during the day (no or yes).
Sleep structure variables | day 1
  Sleep structure was evaluated with the following polysomnography data: sleep onset latency in minutes, rapid eye movement (REM) sleep latency in minutes, wake up after sleep onset (WASO) in minutes, total sleep time in minutes, sleep efficiency (good >85% or bad <84.9%), non-rapid eye movement (NREM) sleep time in stages N1 (%), N2 (%), and N3 (%), rapid eye movement (REM) sleep time (%), arousal, respiratory disturbance index (RDI), index of apnea and hypopnea (IAH).
Sleep Bruxism detection | day 1
  Children and adolescents will be diagnosed with SB, according the criteria of de American Association of Sleep Medicine, if they present: a) regular or frequent tooth grinding sounds occurring during sleep; and b) transient morning jaw muscle pain or fatigue; and/or temporal headache (AASM, 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garg RK, Afifi AM, Garland CB, Sanchez R, Mount DL. Pediatric Obstructive Sleep Apnea: Consensus, Controversy, and Craniofacial Considerations. Plast Reconstr Surg. 2017 Nov;140(5):987-997. doi: 10.1097/PRS.0000000000003752. PMID 29068938
- [Background] Kaditis AG, Alonso Alvarez ML, Boudewyns A, Alexopoulos EI, Ersu R, Joosten K, Larramona H, Miano S, Narang I, Trang H, Tsaoussoglou M, Vandenbussche N, Villa MP, Van Waardenburg D, Weber S, Verhulst S. Obstructive sleep disordered breathing in 2- to 18-year-old children: diagnosis and management. Eur Respir J. 2016 Jan;47(1):69-94. doi: 10.1183/13993003.00385-2015. Epub 2015 Nov 5. PMID 26541535
- [Background] Tan HL, Gozal D, Kheirandish-Gozal L. Obstructive sleep apnea in children: a critical update. Nat Sci Sleep. 2013 Sep 25;5:109-23. doi: 10.2147/NSS.S51907. PMID 24109201
- [Background] Baidas L, Al-Jobair A, Al-Kawari H, AlShehri A, Al-Madani S, Al-Balbeesi H. Prevalence of sleep-disordered breathing and associations with orofacial symptoms among Saudi primary school children. BMC Oral Health. 2019 Mar 12;19(1):43. doi: 10.1186/s12903-019-0735-3. PMID 30866906
- [Background] Andersen IG, Holm JC, Homoe P. Obstructive sleep apnea in children and adolescents with and without obesity. Eur Arch Otorhinolaryngol. 2019 Mar;276(3):871-878. doi: 10.1007/s00405-019-05290-2. Epub 2019 Jan 28. PMID 30689039
- [Background] Baker M, Scott B, Johnson RF, Mitchell RB. Predictors of Obstructive Sleep Apnea Severity in Adolescents. JAMA Otolaryngol Head Neck Surg. 2017 May 1;143(5):494-499. doi: 10.1001/jamaoto.2016.4130. PMID 28241176
- [Background] Chen T, Hughes ME, Wang H, Wang G, Hong X, Liu L, Ji Y, Pearson C, Li S, Hao L, Wang X. Prenatal, Perinatal, and Early Childhood Factors Associated with Childhood Obstructive Sleep Apnea. J Pediatr. 2019 Sep;212:20-27.e10. doi: 10.1016/j.jpeds.2019.05.053. Epub 2019 Jun 26. PMID 31253409
- [Background] Sanchez T, Rojas C, Casals M, Bennett JT, Galvez C, Betancur C, Mesa JT, Brockmann PE. [Prevalence and risk factors for sleep-disordered breathing in chilean schoolchildren]. Rev Chil Pediatr. 2018 Dec;89(6):718-725. doi: 10.4067/S0370-41062018005000902. Spanish. PMID 30725060
- [Background] Krzeski A, Burghard M. Obstructive sleep disordered breathing in children - an important problem in the light of current European guidelines. Otolaryngol Pol. 2018 Jun 29;72(5):9-16. doi: 10.5604/01.3001.0012.1570. PMID 30460910
- [Background] Goyal M, Johnson J. Obstructive Sleep Apnea Diagnosis and Management. Mo Med. 2017 Mar-Apr;114(2):120-124. PMID 30228558
- [Background] Certal V, Catumbela E, Winck JC, Azevedo I, Teixeira-Pinto A, Costa-Pereira A. Clinical assessment of pediatric obstructive sleep apnea: a systematic review and meta-analysis. Laryngoscope. 2012 Sep;122(9):2105-14. doi: 10.1002/lary.23465. Epub 2012 Aug 9. PMID 22886768
- [Background] Brietzke SE, Katz ES, Roberson DW. Can history and physical examination reliably diagnose pediatric obstructive sleep apnea/hypopnea syndrome? A systematic review of the literature. Otolaryngol Head Neck Surg. 2004 Dec;131(6):827-32. doi: 10.1016/j.otohns.2004.07.002. PMID 15577775
- [Background] Abrishami A, Khajehdehi A, Chung F. A systematic review of screening questionnaires for obstructive sleep apnea. Can J Anaesth. 2010 May;57(5):423-38. doi: 10.1007/s12630-010-9280-x. Epub 2010 Feb 9. PMID 20143278
- [Background] De Luca Canto G, Singh V, Major MP, Witmans M, El-Hakim H, Major PW, Flores-Mir C. Diagnostic capability of questionnaires and clinical examinations to assess sleep-disordered breathing in children: a systematic review and meta-analysis. J Am Dent Assoc. 2014 Feb;145(2):165-78. doi: 10.14219/jada.2013.26. PMID 24487608
- [Background] Pabla L, Duffin J, Flood L, Blackmore K. Paediatric obstructive sleep apnoea: can our identification of surgical candidates be evidence-based? J Laryngol Otol. 2018 Apr;132(4):284-292. doi: 10.1017/S0022215118000208. Epub 2018 Feb 14. PMID 29439747